CLINICAL TRIAL: NCT02047305
Title: A Single-center Trial of Endoscopic Radiofrequency Ablation of Moderate and High-grade Intra-epithelial Squamous Neoplasia and Early Flat-type Squamous Cell Carcinoma Using the HALO Ablation System
Brief Title: Radiofrequency Ablation for Patients With Esophageal Squamous Cell Neoplasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Covidien, GI Solutions (Industry)
Responsible Party: Sponsor
Organization: Medtronic - MITG (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B300
Record Dates: First submitted 2014-01-24; First posted 2014-01-28 (Estimated); Results first posted 2020-05-21 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-03

CONDITIONS: ESOPHAGEAL SQUAMOUS CELL CARCINOMA
Keywords: ESCN; RFA
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Radiofrequency ablation (Experimental): To study the safety and effectiveness of radiofrequency ablation (RFA) using the HALO ablation system in completely eradicating the diseased epithelium in patients with ESCN
  Interventions: Device: Radiofrequency Ablation

INTERVENTIONS:
Device: Radiofrequency Ablation — Patients with a histopathological diagnosis of moderate-grade intra-epithelial neoplasia (MGIN), high-grade intra-epithelial neoplasia (HGIN) and/or early flat-type SCCA of the esophagus, are treated with radiofrequency ablation, with repeat endoscopy and follow-up treatment at 3 month intervals.
  Other Names: RFA; Barrx ablation system; HALO ablation system

SUMMARY:
Patients with MGIN, HGIN or flat-type early SCCA of the esophagus will be treated on 3 month intervals with Radiofrequency Ablation (RFA) until complete eradication (CR: no MGIN or worse in the biopsies) will be achieved. All patients will undergo an endoscopy at 12 months after baseline, and the patients with CR will undergo annual endoscopy with biopsies for 5 years.

DETAILED DESCRIPTION:
A patient population with a histopathological diagnosis of moderate-grade intra-epithelial neoplasia (MGIN), high-grade intra-epithelial neoplasia (HGIN) and/or early flat-type SCCA of the esophagus, in lesions measuring 3 to 12cm in length, will be treated with radiofrequency ablation (RFA) using the HALO ablation system. Additional RFA sessions will be performed on 3 month intervals until complete response (CR; no MGIN or worse in biopsies) will be achieved. All patients will then undergo an endoscopy at 12 months after baseline. Patients with CR at 12 months will be followed-up for 5 years with annual endoscopy and biopsies, and additional treatment if necessary. Patients with no CR at 12 months are considered failures.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 18-80 years of age, inclusive
2. Subject meets at least one of the following inclusion criteria:

   1. Within the last 3 months, subject demonstrated a new diagnosis or a reconfirmed diagnosis of squamous MGIN and/or HGIN of the esophagus, or...
   2. within the last 3 months, subject demonstrated a new diagnosis of a flat-type (type 0-IIb) SCCA (G1/G2 only)
3. On endoscopic examination, subject has at least one USL that measures at least 3 cm in at least one dimension and has MGIN or worse (MGIN+) on biopsy
4. The maximum allowable linear length of "USL-bearing esophagus" is 12 cm
5. Baseline EUS (all patients) shows no exclusionary findings for the trial
6. CT scan of chest and upper third of the abdomen (all HGIN and SCCA patients) shows no exclusionary findings for the trial
7. Subject is not pregnant nor has plans to become pregnant in the ensuing 12 months (confirmation of non-pregnant status in women of child-bearing age and ability required with urine or blood test)
8. Subject is eligible for treatment and follow-up endoscopy and biopsy as required by the protocol
9. The subject is willing to provide written, informed consent to participate in this clinical study and understands the responsibilities of trial participation

Exclusion Criteria:

the Eligibility CRF.

1. Esophageal stricture preventing passage of a therapeutic endoscope
2. Any prior endoscopic resection
3. Any esophageal dilation in the past 12 months
4. Any history of a non-squamous cell cancer of the esophagus, or any history of a squamous cell cancer of the esophagus (any stage) prior to 3 months before screening for this trial
5. Any N or M positive status, if patient has a present diagnosis of esophageal SCCA
6. Any previous ablative therapy within the esophagus (photodynamic therapy, multipolar electrical coagulation, argon plasma coagulation, laser treatment, or other) or any radiation therapy to the esophagus.
7. Any previous esophageal surgery, except fundoplication without complications (i.e. no slippage, dysphagia, etc)
8. Evidence of esophageal varices detected within last 6 months or at initial RFA procedure
9. Evidence of eosinophilic esophagitis on endoscopy and/or histology
10. Report of uncontrolled coagulopathy with international normalized ratio (INR) > 2 or platelet count <75,000 platelets per µL (note: a complete blood count is not required for all subjects in this study)
11. Subject is using aspirin, clopidogrel, or non-steroidal anti-inflammatory drugs that can not be discontinued 7 days before and after therapeutic sessions
12. Subject has a known history of unresolved drug or alcohol dependency that would limit ability to comprehend or follow instructions related to informed consent, post-treatment instructions, or follow-up guidelines
13. Subject has an implantable pacing device (examples; AICD, neurostimulator, cardiac pacemaker) and has not received clearance for enrollment in this study by specialist responsible for the pacing device
14. Subject suffers from psychiatric or other illness deemed by the investigator as an inability to comply with protocol
15. Subject has life expectancy less than 2 years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2009-01; Primary Completion 2016-08 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guiqi Wang, MD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] He S, Bergman J, Zhang Y, Weusten B, Xue L, Qin X, Dou L, Liu Y, Fleischer D, Lu N, Dawsey SM, Wang GQ. Endoscopic radiofrequency ablation for early esophageal squamous cell neoplasia: report of safety and effectiveness from a large prospective trial. Endoscopy. 2015 May;47(5):398-408. doi: 10.1055/s-0034-1391285. Epub 2015 Feb 10. PMID 25668428
- [Result] Bergman JJ, Zhang YM, He S, Weusten B, Xue L, Fleischer DE, Lu N, Dawsey SM, Wang GQ. Outcomes from a prospective trial of endoscopic radiofrequency ablation of early squamous cell neoplasia of the esophagus. Gastrointest Endosc. 2011 Dec;74(6):1181-90. doi: 10.1016/j.gie.2011.05.024. Epub 2011 Aug 15. PMID 21839994
- [Derived] Yu X, van Munster SN, Zhang Y, Xue L, Fleischer DE, Weusten BLAM, Lu N, Dawsey SSM, Bergman JJGHM, Wang G. Durability of radiofrequency ablation for treatment of esophageal squamous cell neoplasia: 5-year follow-up of a treated cohort in China. Gastrointest Endosc. 2019 Apr;89(4):736-748.e2. doi: 10.1016/j.gie.2018.10.030. Epub 2018 Oct 26. PMID 30905354

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Radiofrequency Ablation
Started | 96
Completed | 96
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Radiofrequency Ablation
Number analyzed (Participants) | 96
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 59.9 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 52
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Chinese Ethnicity | 96
Region of Enrollment [Number; unit: participants]
  China | 96
Body Mass Index [Mean (Standard Deviation); unit: (kg/m^2)] | 23.4 (2.6)
Current Use of Tabacco [Count of Participants; unit: Participants] | 29
Current Use of Alcohol [Count of Participants; unit: Participants] | 32
History of Cancer [Count of Participants; unit: Participants]
  History of any cancer in a first-degree relative | 29
  Esophageal cancer | 15
Grade of esophageal neoplasia at study entry [Count of Participants; unit: Participants]
  MGIN | 45
  HGIN | 42
  T1m2 ESCC | 9
Length of unstained lesions [Mean (Standard Deviation); unit: CM] | 6.5 (2.9)
Length of treatment area [Mean (Standard Deviation); unit: CM] | 8.6 (2.9)

OUTCOME MEASURES:

1. Primary Outcome: Complete Response
Description: The percentage of subjects demonstrating complete response (CR) defined as complete histological clearance of MGIN, HGIN and SCCA in the treatment area at 12 months after the initial ablation procedure
Time Frame: 12 Month
Measure: Count of Participants; unit: Participants
Arm/Group | Radiofrequency Ablation
Number analyzed (Participants) | 96
Participants | 81

ADVERSE EVENTS:
Arm/Group | Radiofrequency Ablation
All-Cause Mortality (participants affected / at risk) | 0/96
Serious Adverse Events (participants affected / at risk) | 0/96
Other Adverse Events (participants affected / at risk) | 25/96
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Radiofrequency Ablation (N=96)
Mucosal Lacerations (Surgical and medical procedures) | 4
Mucosal Bleb (Surgical and medical procedures) | 1
Stricture (Surgical and medical procedures) | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No